CLINICAL TRIAL: NCT05126017
Title: A Prospective Study to Examine the Validity of a Panel of Objective Burn Scar Measurement Tools
Brief Title: Examine the Validity of a Panel of Objective Burn Scar Measurement Tools
Acronym: BOSS-2
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital Birmingham NHS Foundation Trust (Other)
Collaborators: University of Birmingham (Other); Welsh Burn Centre, Morriston Hospital, Swansea (Unknown); St. Andrews Burn Centre, Broomfield Hospital, Chelmsford (Unknown); The Scar Free Foundation (Unknown)
Responsible Party: Principal Investigator, Naiem Moiemen, Burns and Plastics Consultant, University Hospital Birmingham NHS Foundation Trust
Other Study IDs: RRK7292
Record Dates: First submitted 2021-11-05; First posted 2021-11-18 (Actual); Last update posted 2021-11-18 (Actual); Status verified 2021-11

CONDITIONS: Burns; Scar; Hypertrophic
Keywords: burns; scars; scar assessment; objective assessment; objective scar scale; scar assessment reliability; scar assessment validation
MeSH Terms: conditions — Burns; Cicatrix; Hypertrophy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Bloods and skin biopsy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Reliable scar assessment is essential not only when designing clinical trials to investigate the efficacy of new and existing scar therapies, but also in everyday, clinical practice, to examine the progress of our patients' care. Subjective assessments are extremely important; they demonstrate to the patient the changes and improvements in their scars since the primary burn injury. Nevertheless, clinicians require reliable, validated, and objective tools which can yield measurable and reproducible outcomes. These are ultimately needed to achieve the goal of reducing the physical and psychosocial burden of scarring through compelling research.

Previously, a pilot study (BOSS-1) was conducted in 55 patients with post burn hypertrophic scars. The investigators measured, among other parameters, scar thickness, density, and pliability, using a panel of objective scar assessment tools, alongside standard subjective measurements (questionnaire-based), and skin biopsy assessments. Measurements were performed at a single time point which varied from 3 months to 6 years post burn injury. This work indicated that measuring scar thickness, pliability and colour together, may provide a global scar objective score.

BOSS-2 is a multi-centre study that will validate the preliminary findings in BOSS-1.

DETAILED DESCRIPTION:
The study will recruit 60 burn patients with a burn wound > 1% TBSA that did not achieve 100% wound healing at 3 weeks post injury. Healed wounds will be assessed at 4 time points (3, 12, 18 and 24 months) from time of injury until scar maturation. From the time of recruitment (3 weeks post injury) the open wounds will be closely monitored (clinical assessments, photography and trans-epidermal water loss (TEWL)) until time of complete wound closure will be recorded. The time to healing will be used as a "recognised standard" to validate both the objective and the subjective tools; time to healing has previously been shown to correlate with severity of hypertrophic scarring.

A panel of tools, rather than a single device, has been selected since they capture all scar characteristic changes (thickness, pliability and colour) during the scar maturation process. These objective measurements along with subjective (e.g. POSAS, Vancouver) assessments will be recorded at each time point. At the same time points, blood samples will be taken and 5mm punch biopsy will be taken from SIFTI-2 cohort co-enrolled with BOSS-2 at Queen Elizabeth Hospital Birmingham (QEHB).

The proposed project will: (1) validate the global burn objective scar score, identified in BOSS-1 study; (2) correlate objective versus subjective measures; (3) assess the acceptability of the global scar score with clinicians and patients; (4) correlate the clinical outcomes with tissue and blood scarring markers.

The creation of a validated panel of objective scar measurement devices will form the basis of future scar therapy research (outcome measures for clinical trials). These tools coupled with the haematological and histological data will further the understanding of the process of burn scar maturation and guide future care management.

ELIGIBILITY:
Inclusion Criteria:

* Any individual with burns injury aged ≥ 16 years old.
* Any deep dermal/ full thickness burn but the size must be minimum >1% TBSA
* Patients who can provide informed consent.
* Those treated with split thickness skin grafts or conservatively managed burn wounds which had taken > 3 weeks to heal (<100% healing).

Exclusion Criteria:

* Burns to genitalia, face
* Patients with skin conditions/diseases (pathological fibrosis e.g. scleroderma; pathological thinning e.g. epidermolysis bullosa; collagen disorders e.g. Marfan's syndrome)
* Contraindications to method of scar assessment e.g. known allergy to ultrasound gel
* Chronic steroid use; history of skin malignancy or chronic papulo-squamous disease (e.g. eczema, pemphigus); history of Steven Johnson syndrome/toxic epidermal necrolysis (SJS/TEN) disease
* Patients with history of keloid formation

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All burn patients with burn TBSA >1% deep dermal/full thickness with unhealed burns wounds (<100% healing) at 3 weeks from time of injury.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-01 (Estimated); Primary Completion 2023-08-31 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Global scar score from BOSS-1 | 24 months
  Validate the accuracy of the global scar score that was created in Boss-1 in a larger population sequentially from time of healing to full scar maturation.

SECONDARY OUTCOMES:
Time to 100% healing | 24 months
  Complete wound healing from time of injury
Clinician and patient satisfaction with the various devices | 24 months
  Clinicians and patients will be given a questionnaire at the end of assessments to find out their satisfaction with the devices in terms of comfort, ease of use, and duration.
Correlation of the scores of the objective scar assessment devices to subjective scar measurement scales | 24 months
Early objective global scar score may predict long term outcome | 24 months
Vitamin D | 24 months
Decorin | 24 months
  Immunohistochemistry staining for scar bio-biomarkers including: Decorin
TGF-levels from the serum | 24 months
  Immunohistochemistry staining for scar bio-biomarkers including: Transforming Growth Factor (TGF)

IPD SHARING:
Plan to Share IPD: No